CLINICAL TRIAL: NCT04724421
Title: Expanded Access Protocol for Adults and Pediatric Patients With Sickle Cell Disease Who Have No Alternative Treatment Options
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C534 Expanded Access; C5341025 (Other: Alias Study Number); GBT440-041 (Other: Pfizer); C5341057 (Other: Pfizer)
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Sickle Cell Disease
Keywords: Voxelotor
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Voxelotor — tablet or powder for oral suspension
  Other Names: GBT440

SUMMARY:
The objective of this Expanded Access Protocol (EAP) is to provide voxelotor for the treatment of sickle cell disease (SCD): The study GBT440-041 is the EAP for pediatric patients aged 6 months to 11 years who have no alternative treatment options and are ineligible to participate in a clinical trial of voxelotor and the study C5341057 is the EAP for adults/adolescents 12 years of age and older for patients who cannot satisfactorily be treated with an authorized medicinal product

DETAILED DESCRIPTION:
This EAP may continue until such time that voxelotor is commercially available or the Sponsor discontinues the voxelotor EAP.

Please note that for US sites, enrollment is open only for 6months to < 4 years of age.

ELIGIBILITY:
Inclusion Criteria: GBT440-041

1. Documented diagnosis of sickle cell disease of any genotype
2. Ineligible or unable to participate in actively recruiting clinical studies of voxelotor
3. Baseline hemoglobin (Hb) ≤10.5 g/dL
4. No alternative treatment options in the judgement of the treating Investigator
5. Participants who, if female of childbearing potential (post-menarche), and are sexually active, agree to use highly effective methods of contraception from study start to 30 days after the last dose of voxelotor
6. Written informed parental/guardian consent and participant assent (if applicable) has been obtained per Institutional Review Board (IRB) policy and requirements, consistent with International Council for Harmonisation (ICH) guidelines

Exclusion Criteria: GBT440-041

1. Receiving chronic red blood cell (RBC) transfusion therapy for primary or secondary stroke prevention
2. Hepatic dysfunction characterized by alanine aminotransferase (ALT) >4 × the upper limit of normal (ULN) for age
3. Severe renal dysfunction (estimated glomerular filtration rate [eGFR] <30 mL/min/1.73 m2 by Schwartz formula)
4. Clinically significant bacterial, fungal, parasitic, or viral infection that requires therapy:

   1. Patients with acute bacterial infection requiring antibiotic use should delay screening/enrollment until the course of antibiotic therapy has been completed.
   2. Patients with known active hepatitis A, B, or C or who are known to be Human Immunodeficiency Virus (HIV) positive
5. Any condition affecting drug absorption, such as major surgery involving the stomach or small intestine (prior cholecystectomy is acceptable)
6. Female who is pregnant or breastfeeding
7. Participated in another clinical trial of an investigational drug or medical device, within 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to informed consent for the EAP, or is currently participating in another trial of an investigational drug or medical device
8. Medical, psychological, or behavioral conditions, that, in the opinion of the Investigator, may preclude informed consent, safe participation, or compliance with the protocol procedures
9. Use of herbal medications (eg, St. John's wort), sensitive cytochrome P450 (CYP) 3A4 substrates with a narrow therapeutic index, or strong CYP3A4 inducers
10. Active symptomatic COVID-19 infection

Inclusion Criteria: C5341057

1. Documented diagnosis of SCD of any genotype confirmed by laboratory genetic testing
2. Aged 12 years and older
3. Haemoglobin ≥5.5 and ≤ 10.5 g/dL, based on a test performed according to local standard of care
4. Patient cannot be treated satisfactorily with any authorised medicinal product
5. Patient or their legal representative has provided written informed consent to participate in the voxelotor EAP for the treatment of SCD
6. Patient or their legal representative has provided written informed consent on data processing and protection

Exclusion Criteria: C5341057

1. Patients with clinically significant bacterial, fungal, parasitic or viral infection which requires therapy.
2. History of serious drug hypersensitivity reaction to voxelotor or excipients
3. Participated in another clinical trial of an investigational agent (or medical device) within 30 days of participation in EAP.
4. Medical, psychological, or behavioral condition that, in the opinion of the study doctor, would confound or interfere with evaluation of safety and/or effectiveness of the study drug, prevent compliance with the study protocol; preclude informed consent; or render the participant unable/unlikely to comply with the study procedures

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (33):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Rady Children's Hospital San Diego, San Diego, California
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Hospital / Children's National Health System, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Baptist Medical Center/Wolfson Children's Hospital, Jacksonville, Florida
  - Nemours Children's Health, Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Children's Healthcare of Atlanta Scottish Rite, Atlanta, Georgia
  - AU Medical Center Clinical Research Pharmacy, Augusta, Georgia
  - Augusta University, Augusta, Georgia
  - Children's Hospital of Georgia, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Tulane Lakeside, Metairie, Louisiana
  - Tulane University Hospitals and Clinics, New Orleans, Louisiana
  - Children's Hospital, New Orleans, Louisiana
  - Childrens Hospital of NOLA, New Orleans, Louisiana
  - University Of Michigan Hospitals, Ann Arbor, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center & Children's Hospital of New Jersey, Newark, New Jersey
  - BronxCare Health System, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - East Carolina University Brody School of Medicine(ECU), Greenville, North Carolina
  - ECU Physicians, Brody Outpatient Clinic, Greenville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Medical University of South Carolina: Investigational Drug Services Pharmacy, Charleston, South Carolina
  - Medical University of South Carolina: Shawn Jenkins Women's and Children's Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health - Upstate, Greenville, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Health Care System, Fort Worth, Texas
  - Pediatric Specialists of Virginia (Inova Ashburn HealthPlex), Ashburn, Virginia
  - Pediatric Specialists of Virginia (Schar Cancer Institute), Fairfax, Virginia
- Brazil (4):
  - Multihemo Serviços Médicos S/A, Recife, Pernambuco
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo
  - HEMORIO - Hematologia Laboratorial, Rio de Janeiro
  - ESHO Empresa de Serviços Hospitalares S.A/ Hospital Samaritano de Higienópolis, São Paulo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-041